CLINICAL TRIAL: NCT07399145
Title: Comparison of the Effects of Prolotherapy and Rehabilitation Treatments in Low Back Pain
Brief Title: Comparison of Prolotherapy and Rehabilitation Treatments in Low Back Pain (CPRTLBP)
Acronym: CPRTLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balnear and Rehabilitation Sanatorium Techirghiol (Other)
Responsible Party: Principal Investigator, Elena-Valentina Ionescu, Professor (Associate) Dr. Ionescu Elena Valentina, Balnear and Rehabilitation Sanatorium Techirghiol
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StelianMociu
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Low Back Pain
Keywords: chronic low back pain; physiotherapy; balneotherapy; prolotherapy; pain assessment; functional disability; quality of life
MeSH Terms: conditions — Low Back Pain | interventions — Prolotherapy; Balneology; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolotherapy group (PG) (Experimental): The prolotherapy intervention was delivered over three sessions, performed at three-week intervals. All procedures were performed bilaterally under continuous ultrasound guidance using a BK Medical Flex Focus 800 ultrasound system with a convex probe.
  The prolotherapy solution was administered at predefined anatomical sites identified sonographically, including one injection point corresponding to the piriformis muscle, five points along the iliac crests corresponding to ligamentous insertions, three points at the sacral level, and five points at the level of the lumbar transverse processes targeting paravertebral ligamentous insertions. In addition, five unilateral injections were performed at the level of the lumbar spinous processes. In total, 33 injection points were used per session.
  Interventions: Other: Prolotherapy
- Balneotherapy plus Physiotherapy Group (BG) (Experimental): Participants assigned to the balneotherapy group (BG) completed a structured two-week inpatient rehabilitation program comprising 10 treatment days at the Balneal and Rehabilitation Sanatorium Techirghiol, Romania.
  Interventions: Other: Balneotherapy plus Physiotherapy
- Physiotherapy Control Group (CG) (Active Comparator): Participants allocated to the control group (CG) were assessed and managed at the Ovidius Clinical Hospital in Romania, where they received a conventional conservative treatment program.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Prolotherapy — A volume of 1 mL of prolotherapy solution was administered at each injection site. The injected solution consisted of a 1:1 dilution of 33% dextrose and 1% lidocaine, resulting in a final dextrose concentration of 16.5%. This formulation was used consistently across all injection sites to ensure standardized delivery and reproducibility of the therapeutic effect. All infiltration procedures were performed under strict aseptic conditions. The interventions were conducted under intravenous analgosedation, using a single-dose regimen of midazolam (2 mg), propofol (approximately 60 mg), and fentanyl (0.1 mg), administered to ensure patient comfort and procedural compliance. After each treatment session, patients were observed clinically to monitor for any immediate adverse events or procedure-related complications.
  Arms: Prolotherapy group (PG)
Other: Balneotherapy plus Physiotherapy — The intervention was based on the region's specific natural therapeutic resources and was conducted under continuous medical supervision. The treatment schedule included saline therapeutic pool baths combined with supervised exercise therapy and applications of sapropelic therapeutic mud, with sessions performed daily, five days per week.
  Alongside balneological treatments, patients received daily electrotherapy following a standardized protocol, which consisted of lumbar magnetotherapy, interferential current therapy, and therapeutic ultrasound.
  The rehabilitation program also incorporated daily massage therapy and supervised therapeutic exercises carried out in a dedicated rehabilitation gym.
  Arms: Balneotherapy plus Physiotherapy Group (BG)
Other: Physiotherapy — The therapeutic program consisted of physiotherapy combined with structured exercise therapy targeting lumbar spine stabilization and mobility, along with electrotherapy and massage therapy. No balneological interventions or prolotherapy procedures were included in the management of this group.
  Arms: Physiotherapy Control Group (CG)

SUMMARY:
Chronic low back pain (CLBP) represents one of the leading causes of long-term disability among adults and places a substantial strain on healthcare systems globally. The clinical course of CLBP is highly heterogeneous, with considerable variability in symptom persistence and functional impairment, which complicates therapeutic decision-making in routine practice.

Conventional physiotherapy is commonly prescribed for patients with CLBP; however, evidence comparing its short-term effectiveness with alternative interventions such as balneotherapy and prolotherapy remains scarce. Balneotherapy, often used as an adjunct to physiotherapy, is widely applied in the management of chronic musculoskeletal conditions and is believed to provide therapeutic benefits through a combination of thermal and mechanical effects.

In addition, psychosocial factors play a crucial role in the evolution of low back pain. Increased stress, insufficient social support, occupational dissatisfaction, and mood disorders have been associated with a higher likelihood of pain chronicification and reduced response to treatment.

The objective of the present study was to evaluate and compare short-term clinical outcomes of standard physiotherapy, combined balneotherapy and physiotherapy, and prolotherapy in individuals with chronic low back pain. Outcomes were assessed using validated instruments measuring pain severity, functional disability, lumbar spine mobility, quality of life, and psychological well-being at baseline and after a four-week intervention period.

The study enrolled adults aged 18 to 70 years with CLBP persisting for more than three months and a baseline Visual Analog Scale (VAS) score of at least 4. Participants were assigned to one of three treatment modalities: physiotherapy alone, balneotherapy combined with physiotherapy, or prolotherapy. Participants allocated to the dextrose prolotherapy group (PG) and the standard physiotherapy control group (CG) were treated at Ovidius Clinical Hospital, Romania, while patients included in the balneotherapy plus physiotherapy group (BG) underwent treatment at the Balneal and Rehabilitation Sanatorium Techirghiol, Romania. Evaluations were conducted at baseline (T0) and at the four-week follow-up (T1), encompassing measures of pain intensity, functional limitation, lumbar mobility, quality of life, and psychological status.

The results highlight the potential benefits of multimodal and regenerative therapeutic approaches within personalized conservative treatment strategies for patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CLBP lasting more than three months, confirmed by lumbar radiography or magnetic resonance imaging
* Pain intensity of at least 4 on the Visual Analog Scale
* Age between 18 and 70 years
* Patients who can comply with the study protocol and scheduled evaluations
* Patients who provided written informed consent before participation

Exclusion Criteria:

* Lumbar disc herniation with surgical indication or severe radiculopathy
* Active infections
* Systemic inflammatory or autoimmune diseases
* A history of allergy to substances used in dextrose prolotherapy
* Contraindications to balneotherapy, such as severe cardiovascular disease, renal insufficiency, or severe dermatological conditions
* Prior prolotherapy or balneotherapy within six months before enrollment
* Decompensated chronic cardiovascular, hepatic, renal, respiratory, or neurological diseases at the time of inclusion
* Pregnancy
* Breastfeeding
* Active neoplastic disease
* Decompensated psychiatric disorders
* Allergies to natural therapeutic factors that could lead to treatment interruption
* Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline and follow-up assessments were conducted at 4 weeks after treatment completion
  Pain intensity was assessed using the Visual Analog Scale (VAS). Participants were asked to rate their current pain intensity by marking a point on a 100-mm horizontal line, where 0 indicates "no pain", and 100 indicates "worst pain imaginable." The score was recorded in millimeters (mm). Outcome range and interpretation: Minimum value: 0, Maximum value: 100. Higher scores indicate worse pain intensity.

SECONDARY OUTCOMES:
Functional disability | Baseline and follow-up assessments were conducted at 4 weeks after treatment completion
  Functional disability was assessed using the Roland-Morris Disability Questionnaire (RMDQ). The questionnaire consists of 24 items related to physical activities and daily functioning affected by low back pain. Participants were asked to mark each statement that applied to their condition on the day of assessment. Each marked item was scored 1 point, and unmarked items were scored 0 points. The total score was calculated by summing all marked items and is reported as a unitless score. Outcome range and interpretation: Minimum value: 0, Maximum value: 24. Higher scores indicate greater functional disability (worse outcome), while lower scores indicate less disability (better outcome).
Lumbar spine mobility | Baseline and follow-up assessments were conducted at 4 weeks after treatment completion
  Lumbar spine mobility was assessed using the Schober test. With the participant standing upright, a point was marked at the level of the lumbosacral junction (L5-S1), and a second point was marked 10 cm above the first mark. Participants were then asked to bend forward maximally, and the distance between the two marks was remeasured. The increase in distance during trunk flexion was recorded in centimeters (cm) and used as the measure of lumbar spine mobility. Outcome range and interpretation: Minimum value: 0 cm, Maximum value: depending on individual mobility. Higher values indicate greater lumbar spine mobility (better outcome), while lower values indicate reduced mobility (worse outcome).
Psychological status | Baseline and follow-up assessments were conducted at 4 weeks after treatment completion
  Psychological status was assessed using the Hospital Anxiety and Depression Scale (HADS), which consists of 14 items divided into two subscales: anxiety (HADS-A) and depression (HADS-D), each containing 7 items. Participants were asked to rate how they had been feeling over the previous week. Each item is scored on a 4-point Likert scale ranging from 0 to 3. Subscale scores were calculated by summing the relevant item scores and are reported as unitless scores.Outcome range and interpretation: HADS-A (Anxiety): Minimum value: 0, Maximum value: 21. Higher scores indicate greater anxiety severity (worse psychological status). HADS-D (Depression): Minimum value: 0, Maximum value: 21. Higher scores indicate greater depressive symptom severity (worse psychological status).

CONTACTS AND LOCATIONS:
Locations (1):
- Balneal and Rehabilitation Sanatorium of Techirghiol, Constanța, Techirghiol, Romania

REFERENCES:
- [Background] Antonelli M, Donelli D, Veronesi L, Vitale M, Pasquarella C. Clinical efficacy of medical hydrology: an umbrella review. Int J Biometeorol. 2021 Oct;65(10):1597-1614. doi: 10.1007/s00484-021-02133-w. Epub 2021 Apr 17. PMID 33866427
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] Anheyer D, Klose P, Koch AK, Haller H, Dobos G, Cramer H. Comparative efficacy of different exercise interventions in chronic non-specific low back pain: protocol of a systematic review and network meta-analysis. BMJ Open. 2020 Aug 5;10(8):e036050. doi: 10.1136/bmjopen-2019-036050. PMID 32759244
- [Background] Linton SJ. A review of psychological risk factors in back and neck pain. Spine (Phila Pa 1976). 2000 May 1;25(9):1148-56. doi: 10.1097/00007632-200005010-00017. PMID 10788861
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Goodman A, Bell DA, Rice LW. DNA ploidy status: its impact on early-stage endometrial adenocarcinoma. Gynecol Oncol. 1993 Dec;51(3):355-61. doi: 10.1006/gyno.1993.1303. PMID 8112645